CLINICAL TRIAL: NCT07302139
Title: Risk of Metachronous Advanced Colorectal Neoplastic Among Individuals With Varying Numbers of Non-Advanced Adenomas Detected During Screening Colonoscopy: A Retrospective Observational Study
Brief Title: Risk of Metachronous Advanced Colorectal Neoplastic Among Individuals With Varying Numbers of Non-Advanced Adenomas Detected During Screening Colonoscopy
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Other Study IDs: 2025K369
Record Dates: First submitted 2025-11-29; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Adenoma
Keywords: Screening colonoscopy; Surveillance; Advanced colorectal adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Individuals with <3 NAAs detected during screening colonoscopy: Individuals with <3 non-advanced adenomas detected during screening colonoscopy
  Interventions: Other: No Intervention: Observational Cohort
- Individuals with 3-4 NAAs detected during screening colonoscopy: Individuals with 3-4 non-advanced adenomas detected during screening colonoscopy
  Interventions: Other: No Intervention: Observational Cohort
- Individuals with >4 NAAs detected during screening colonoscopy: Individuals with >4 non-advanced adenomas detected during screening colonoscopy
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention: Observational Cohort

SUMMARY:
A retrospective observational study to evaluate the risk of metachronous advanced colorectal neoplastic (ACRN) among individuals with varying numbers of non-advanced adenomas (NAA) detected during screening colonoscopy

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most commonly diagnosed malignancy worldwide and the second leading cause of cancer-related mortality. In recent years, with increasing westernization of diet and lifestyle, both the incidence and prevalence of CRC in China have risen sharply. CRC has become the most common gastrointestinal malignancy in the country, ranking second in incidence and fifth in mortality among all cancers. Screening colonoscopy and appropriate surveillance intervals can substantially reduce CRC-related deaths.

The latest 2020 U.S. Multi-Society Task Force (USMSTF) guidelines classify patients with 1-2 non-advanced adenomas (NAAs), 3-4 NAAs, and >4 NAAs as having low-, intermediate-, and high-risk colonoscopic findings, respectively, and recommend surveillance intervals of 7-10 years, 3-5 years, and 3 years for these groups. However, accumulating evidence suggests that the risk of developing metachronous advanced colorectal neoplastic lesions (ACRN) in individuals with 3-4 NAAs may be comparable to those with only 1-2 NAAs, raising concerns regarding the appropriateness of current surveillance recommendations.

Using a real-world, endoscopy database, this study systematically evaluates the association between different NAA counts and the subsequent risk of ACRN, providing evidence to inform optimization of post-polypectomy surveillance intervals.

ELIGIBILITY:
Inclusion Criteria:

* First-time screening colonoscopy
* Only non-advanced adenomas (no villous features, no high-grade dysplasia, and diameter <10 mm) were detected during first-time screening colonoscopy
* Individuals with at least one surveillance colonoscopy
* Complete electronic medical record and pathology information

Exclusion Criteria:

* Inadequate bowel preparation (BBPS < 6)
* Emergency colonoscopy
* History of colorectal cancer
* Incomplete pathology information or incompletely resected polyps
* Screening colonoscopies performed by endoscopists with a low dynamic adenoma detection rate (ADR < 15%)
* Follow-up duration < 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who underwent their first-time screening colonoscopy between 2012 and 2023 at the endoscopy centers of Huadong Hospital and Shanghai Tongji Hospital, and who completed at least one surveillance colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 2955 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Metachronous Advanced Colorectal Neoplasia | Through study completion, an average of 1 month
  Metachronous advanced colorectal neoplasia is defined as advanced adenoma (≥10 mm, villous component, or high-grade dysplasia) or colorectal cancer detected at any follow-up colonoscopy after the baseline index colonoscopy.

SECONDARY OUTCOMES:
Incidence of Metachronous Colorectal Neoplasia | Through study completion, an average of 1 month
  Metachronous colorectal neoplasia is defined as any adenoma or colorectal cancer detected at any follow-up colonoscopy after the baseline index colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Danian Ji, M.D., Study Director — Huadong Hospital
Locations (1):
- Huadong hospital, Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after completion of this study
Access Criteria: All researchers can require the original data from principal investigator of this study (Email address: arctg4@163.com)